CLINICAL TRIAL: NCT02639975
Title: Randomized, Double Blind, Placebo Controlled "First-in-human" Study To Assess the Safety and Tolerability of Single Ascending Oral Doses of PBF-677 ( 100 mg, 200 mg, 400 mg and 600 mg ) in Healthy Young Male Volunteers
Brief Title: "First-in-human" Study To Assess the Safety and Tolerability of PBF-677 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Palobiofarma SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CUNFI-1509
Record Dates: First submitted 2015-12-17; First posted 2015-12-28 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2016-09

CONDITIONS: Glaucoma
Keywords: Adenosine A3 receptor antagonist
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 100 mg PBF-677 (Experimental)
  Interventions: Drug: PBF-677
- 200 mg PBF-677 (Experimental)
  Interventions: Drug: PBF-677
- 400 mg PBF-677 (Experimental)
  Interventions: Drug: PBF-677
- 600 mg PBF-677 (Experimental)
  Interventions: Drug: PBF-677
- Placebo 100 mg (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo 200 mg (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo 400 mg (Placebo Comparator)
  Interventions: Drug: Placebo
- Placebo 600 mg (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PBF-677 — once daily oral administration
  Arms: 100 mg PBF-677; 200 mg PBF-677; 400 mg PBF-677; 600 mg PBF-677
Drug: Placebo — once daily oral administration
  Arms: Placebo 100 mg; Placebo 200 mg; Placebo 400 mg; Placebo 600 mg

SUMMARY:
The proposed trial a "Randomized, Double Blind, Placebo Controlled "first in-human" Study to Assess the Safety and Tolerability of Single Ascending Oral Doses of PBF-677 in Male Healthy Volunteers" (Protocol Code No:CUNFI-1509 EudraCT No:2015-003546-57) will be a single-centre, randomized, double-blind, dose escalation study without therapeutic benefit, in which PBF-677 will be administered as single, oral, ascending-dose to volunteers.

Up to four different rising doses (100 mg, 200 mg, 400 mg and 600 mg) will be tested in groups of 8 participants; in each dose level participants will be randomized to active drug or placebo in a 6:2 fashion. As this will be the first time that PBF-677 in going to be administered to humans, as a safety measure a stepwise drug administration will be performed in each cohort. The volunteers of each cohort will be divided in 3 blocks/subgroups: Initially, one volunteer will receive active drug (subgroup 1). After 48h of safety and tolerability assessment, a second subgroup of 3 volunteers will receive 2 active drug and 1 placebo and after further 48h of safety and tolerability assessments a third subgroup of 4 volunteers will receive 3 active drug and 1 placebo. After evaluation of safety, parameters of corresponding dose level the process will replicate one week afterwards in the following dosages.

The principal variable safety and tolerability of PBF-677 will be evaluated with physical records (Electrocardiogram (ECG), vital signs, blood chemistry and haematology, conducted before, during and after study course). Assessment of the pharmacokinetic profile (Maximum plasma concentration of the drug (peak) after single dose (Cmax),Time necessary to reach Cmax (tmax), Area under the time-concentration curve to "zero" to time "t" (AUC0t), and Elimination half-life (t1/2) of PBF-677 will be included as secondary variable.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects, 18-45 years (inclusive) of age at the time of enrollment.
2. Males should agree to abstain from sexual intercourse with a female partner or agree to use a condom with spermicide, in addition to having their female partner use some contraceptive measures as oral contraceptive drugs, intrauterine hormonal contraception, or cervical caps until 28 days post-administration.
3. Clinically acceptable blood pressure and pulse rate in supine and standing position (SBP between 140-100 mm Hg/ DBP between 90-50 mm Hg / HR between 100-50 bpm). Blood pressure and pulse will be measured after a minimum of 3 minutes of resting.
4. Body weight within normal range (Quetelet's index between 19 and 26) expressed as weight (kg) / height (m2).
5. Able to understand the nature of the study and comply with all their requirements.
6. Free acceptance to participate in the study by obtains signed informed consent form approved by the Ethics Committee (CEIC).

Exclusion Criteria:

1. History of serious adverse reactions or hypersensitivity to any drug.
2. Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
3. Background or clinical evidence of chronic diseases.
4. Acute illness two weeks before drug administration.
5. Having undergone major surgery during the previous 6 months.
6. Smokers (refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc., for 6 months prior to the administration of the study medication).
7. History of alcohol dependence or drug abuse in the last 5 years or daily consumption of alcohol > 40 g or high consumption of stimulating beverages (> 5 coffees, teas or coca cola drinks/ day).
8. Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
9. Need of any prescription medication within 14 days prior to the administration of the investigational drug and non prescription medication or herbal medicines within 7 days prior to the administration of the drug. Paracetamol (acetaminophen) is allowed, at doses up to 1 g daily, at the investigator discretion.
10. Participation in other clinical trials during the previous 90 days in which an investigational drug or a commercially available drug was tested.
11. Having donated blood during 3 months period before inclusion in the study.
12. Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e. impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhea or conditions associated with total or partial obstruction of the urinary tract
13. 12 lead ECG obtained at screening with PR ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec, bradycardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval.
14. Symptoms of a significant somatic or mental illness in the four week period preceding drug administration.
15. History of hepatitis HBV and / or HCV and / or positive serology results which indicate the presence of hepatitis B surface antigen and / or detectable HCV ribonucleic acid (RNA).
16. Positive results from the HIV serology.
17. Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening evaluation.
18. Positive results of the drugs at screening period or the day before starting treatment period. A minimum list of 6 drugs will be screened for inclusion: Amphetamines, Cocaine, Ethanol, Opiates, Cannabinoids and Benzodiazepines (positive results may be repeated at the discretion of the Principal Investigator).
19. Known hypersensitivity to the study drug or the composition of the galenical form.
20. History of psychiatric diseases or epileptic seizures.
21. Pill swallowing difficulties.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events | 1 week
  The occurrence of adverse events will be monitored through the complete study. Adverse events will be recorded with the following information: severity grade (mild, moderate, severe); suspected/unsuspected relationship to the study drug; duration (date and time of onset, defined as precisely as possible, and end date or if continuing at final exam)

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values | 5-7 days post administration
  The following laboratory evaluations will be performed at the study site:
  * Hematology - Hemoglobin, Hematocrit, White Blood Cells (WBC) with differential, Red Blood Cells (RBC) count, Platelet count.
  * Biochemistry - Sodium, Potassium, Calcium, Inorganic Phosphorus, Total Proteins, Total Bilirubin, Albumin, Fasting Cholesterol, Fasting Triglycerides, Serum Creatinine, Creatine Kinase (CK), Fasting Glucose, Aspartate amino transferase (AST), Alanine amino transferase (ALT), Glutamyl transpeptidase (GGT), Alkaline Phosphatase, BUN (urea-N), Uric Acid.
  * Urinalysis - Glucose, Leukocytes, Ketonic Bodies, Nitrites, Proteins, Bilirubin, Urobilinogen and Erythrocytes. A midstream urine sample will be obtained, in order to avoid contamination and allow a proper assessment.
Electrocardiogram (EKG) | [pre-dose], [+ 40min], [+ 1.5h], [+ 3h], [+ 24h] and Days (5-7) post-medication
Vital signs | [pre-dose], [+ 20 min], [+ 60min], [+ 2h], [+ 4h], [+ 8h], [+ 12h] , [+ 24h] and Days (5-7) post-medication
  This evaluation will include automated/manual assessments of systolic and diastolic blood pressure, heart and respiratory rate.
Physical examination | At day-1 (predose), at + 24h post-drug administration and at the follow-up (5-7) days
  This evaluation will include an examination of general appearance, eyes, throat-nose-ears, teeth, skin, lung, heart, abdomen general, liver, spleen, kidneys, spine, lymph nodes, extremities, short neurological status. Genital, urinary tract and rectal examination will not be done on a routine basis.
Maximum plasma concentration of PBF-677 (peak) after single dose (Cmax) | 0-24 h post dose
  The Blood extractions will be done at the following time points: Baseline [pre-dose], [+ 10 min], [+ 20 min], [+ 40 min], [+ 60 min], [+ 1.5h], [+ 2 h], [+ 2.5 h], [+ 3 h], [+ 4h], [+ 8h], [+ 12h], [+16h] and [+ 24h] post-medication. Plasma concentrations of parent compound (PBF-677) will be measured with a previously validated method. The Pharmacokinetic (PK) parameter will be derived from each individual plasma concentration versus time profile using standard methods.
Time necessary to reach Maximum plasma concentration of PBF-677 (Tmax) | 0-24 h post dose
  The Blood extractions will be done at the following time points: Baseline [pre-dose], [+ 10 min], [+ 20 min], [+ 40 min], [+ 60 min], [+ 1.5h], [+ 2 h], [+ 2.5 h], [+ 3 h], [+ 4h], [+ 8h], [+ 12h], [+16h] and [+ 24h] post-medication. Plasma concentrations of parent compound (PBF-677) will be measured with a previously validated method. The Pharmacokinetic (PK) parameter will be derived from each individual plasma concentration versus time profile using standard methods.
Area under the time-concentration curve to "zero" to time "t" (AUC0t) | 0-24 h post dose
  The Blood extractions will be done at the following time points: Baseline [pre-dose], [+ 10 min], [+ 20 min], [+ 40 min], [+ 60 min], [+ 1.5h], [+ 2 h], [+ 2.5 h], [+ 3 h], [+ 4h], [+ 8h], [+ 12h], [+16h] and [+ 24h] post-medication. Plasma concentrations of parent compound (PBF-677) will be measured with a previously validated method. The Pharmacokinetic (PK) parameter will be derived from each individual plasma concentration versus time profile using standard methods.
Elimination half-life (t1/2) of PBF-677 | 0-24 h post dose
  The Blood extractions will be done at the following time points: Baseline [pre-dose], [+ 10 min], [+ 20 min], [+ 40 min], [+ 60 min], [+ 1.5h], [+ 2 h], [+ 2.5 h], [+ 3 h], [+ 4h], [+ 8h], [+ 12h], [+16h] and [+ 24h] post-medication. Plasma concentrations of parent compound (PBF-677) will be measured with a previously validated method. The Pharmacokinetic (PK) parameter will be derived from each individual plasma concentration versus time profile using standard methods.